CLINICAL TRIAL: NCT00596323
Title: Implantable Antenna Sensors for Continuous Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Elaine Moreland MD, UAB
Other Study IDs: X070207013
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: antenna; continuous glucose monitoring; electromagnetic
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The researchers' long-term goal is to develop a small implantable device that can continually monitor glucose levels. This will be an antenna. Changes in the glucose levels in will affect the antenna signals and those can be used to predict the patient's glucose levels.

DETAILED DESCRIPTION:
Our goal is to develop a small size implantable device that can continually monitor glucose levels. The scientific objective of this application is to examine the efficacy of using implantable antennas to measure the glucose levels. The central hypothesis of this application is that the changes in the glucose levels in the medium surrounding the antenna will affect the antenna parameters such as input impedance and resonance frequency, and these changes can be used to predict the patient's glucose levels. We have formulated this hypothesis on the basis of our preliminary data, which will be detailed later, in the Preliminary Studies section. The rationale for the proposed research is that, once the correlation between the glucose levels and antenna parameters are determined, the design of a miniaturized long term glucose monitoring device will become a reality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult able to give a blood sample

Exclusion Criteria:

* Adults with diabetes or other glycemic or hematologic disorders.
* Sick adults

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Moreland, MD, Study Director — University of Alabama at Birmingham
Locations (1):
- University of Alabama Children's Hospital, Birmingham, Alabama, United States